CLINICAL TRIAL: NCT02510911
Title: Does Caffeine Reduce Postoperative Bowel Paralysis After Elective Colectomy? - A Randomized, Placebo-controlled Trial
Brief Title: Does Caffeine Reduce Postoperative Bowel Paralysis After Elective Colectomy?
Acronym: CaCo
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of effect at interims analysis
Sponsor: Thomas Steffen (Other)
Collaborators: Gottfried und Julia Bangerter- Rhyner-Stiftung, Basel (Other)
Responsible Party: Sponsor-Investigator, Thomas Steffen, Deputy head of department, Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CaCo, Chir201401
Record Dates: First submitted 2015-07-27; First posted 2015-07-29 (Estimated); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Postoperative Ileus; Laparoscopic Colectomy Without Stoma Formation; Colorectal Neoplasm; Diverticulitis
Keywords: colectomy; laparoscopy; caffeine
MeSH Terms: conditions — Colorectal Neoplasms; Diverticulitis | interventions — Caffeine; Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Caffeine (100 mg) (Experimental): Verum 1 with 100 mg caffeine
  Interventions: Drug: Caffeine (100 mg); Other: Radiopaque marker
- Caffeine (200 mg) (Experimental): Verum 2 with 200 mg caffeine
  Interventions: Drug: Caffeine (200 mg); Other: Radiopaque marker
- corn starch (250 mg approx.) (Placebo Comparator): approx. 250 mg corn starch as placebo
  Interventions: Drug: corn starch (250 mg approx.); Other: Radiopaque marker

INTERVENTIONS:
Drug: Caffeine (100 mg) — Patients after laparoscopic colectomy will receive 3 times daily capsules with 100 mg caffeine together with the meals.
  First capsule will be taken on the evening of surgery if surgery was completed before 1 pm, otherwise the first capsule will be taken on the morning of the next day.
  Treatment consists of 10 capsules and will be stopped after the first solid bowel movement.
  Other Names: coffeinum; methyltheobromine; 1,3,7-trimethyl-3,7-dihydro-1H-purin-2,4-dion; CAS No: 56-08-2; Ph.Eur: 6.0/027; ATC code: N06BC01
  Arms: Caffeine (100 mg)
Drug: Caffeine (200 mg) — Patients after laparoscopic colectomy will receive 3 times daily capsules with 200 mg caffeine together with the meals.
  First capsule will be taken on the evening of surgery if surgery was completed before 1 pm, otherwise the first capsule will be taken on the morning of the next day.
  Treatment consists of 10 capsules and will be stopped after the first solid bowel movement.
  Other Names: coffeinum; methyltheobromine; 1,3,7-trimethyl-3,7-dihydro-1H-purin-2,4-dion; CAS No: 56-08-2; Ph.Eur: 6.0/027; ATC code: N06BC01
  Arms: Caffeine (200 mg)
Drug: corn starch (250 mg approx.) — Patients after laparoscopic colectomy will receive 3 times daily capsules with 250 mg corn starch together with the meals.
  First capsule will be taken on the evening of surgery if surgery was completed before 1 pm, otherwise the first capsule will be taken on the morning of the next day.
  Treatment consists of 10 capsules and will be stopped after the first solid bowel movement.
  Other Names: Amylum maydis
  Arms: corn starch (250 mg approx.)
Other: Radiopaque marker — On the morning of the first, second and third day after surgery patients will take 1 capsule each day with radiopaque markers .
  On day 4 after surgery an abdominal X-ray will be performed to localize the markers.
  Each gelatin capsule contains 10 markers consisting of polyurethane encapsulated barium sulfate (40%).
  Other Names: Colon Transit; PZN 3351272; GTIN Code 7629999004153

SUMMARY:
Postoperative bowel paralysis is common after abdominal operations, including colectomy. As a result, hospitalization may be prolonged leading to increased cost. A recent randomized controlled trial from the University of Heidelberg showed that consumption of regular black coffee after colectomy is safe and associated with a significantly faster resumption of intestinal motility (Müller 2012). The mechanism how coffee stimulates intestinal motility is unknown but caffeine seems to be the most likely stimulating agent.

Thus, this trial addresses the question: Does caffeine reduce postoperative bowel paralysis after elective laparoscopic colectomy?

Patients after laparoscopic colectomy will receive either 100 mg caffeine, 200 mg caffeine, or 250mg corn starch (placebo) 3 times daily in identically looking gelatin capsules.

The study is a randomized, controlled trial, with blinding of physicians, patients and nursing stuff (evaluating the endpoints).

Primary endpoint will be the time to first bowel movement.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective laparoscopic colectomy (right or left hemicolectomy, segmental resection, extended hemicolectomy, sigmoid resection, upper rectum (anastomosis higher than 7 cm ab ano))
* There will be no upper age limit. If elderly patients are considered fit for surgery, they will be included in the study.
* Informed consent
* Application of epidural analgesia

Exclusion Criteria:

* Participation in another concurrent interventional trial
* Need for a stoma (colostomy or ileostomy) or reversal of a stoma, if the patient had a complete bowel obstruction
* Known hypersensitivity or allergy to caffeine/coffee
* Expected lack of compliance
* American Society of Anesthesiologists (ASA) Physical Status Score of IV or V
* Impaired mental state or language problems
* Alcoholism or drug abuse
* Previous extensive abdominal surgery
* Inflammatory bowel disease
* Clinically significant cardiac arrhythmia
* Cardiac insufficiency
* Pregnancy, lactation, or childbearing potential without using adequate contraception
* Intake of opioid analgesics, or steroids >5mg/d for ≥7 days before surgery
* Under anti-depressive medication
* Liver cirrhosis or compromised liver function (MELD score >15)
* Emergency procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-08; Primary Completion 2020-08 (Actual); Study Completion 2020-12-22 (Actual)

PRIMARY OUTCOMES:
Time to first bowel movement | 7 days
  Time from end of surgery (time of closing suture) until patient's first bowel movement (passage of stool) in hours.
  A patient is considered to have met the primary endpoint when he or she had first tolerated food (recovery of upper GI function) and experienced a bowel movement for the first time (recovery of lower GI function).

SECONDARY OUTCOMES:
Time to first flatus | 7 days
  Time from end of surgery until patient's first flatus in hours. The passage of flatus will be determined by questioning the patient; the passage of a bowel movement will be determined by reference to nursing records or by the clinical judgment of the investigator or designee following questioning the patient.
Time to tolerance of solid food | 7 days
  Time from end of surgery until patient tolerates intake of solid food in hours. Tolerance of food is defined as the first time the patient is able to eat solid food (any food re-quiring chewing) without vomiting or significant nausea within 4 h after the meal, and without reversion to only enteral fluids.
Postoperative vomiting events | 7 days
  Number of times patient has to vomit.
Colonic passage time | 4 days
  On day 1, 2 and 3 after surgery patients take one capsule with radioopaque markers. On day 4 location and count of markers is determined by X-ray imaging and the colonic passage time is determined (Metcalf 1987).
Actual postoperative hospital stay | 30 days
  Number of days from surgery until actual discharge.
Theoretical postoperative hospital stay | 30 days
  Days from surgery until patient would be fit for release. Often patients stay longer in hospital than clinically required. Thus, evaluation of theoretical hospital stay.
  A patient is fit for release if:
  * there had been bowel movement
  * solid food is tolerated
  * no serious pain
  * unproblematic mobilisation
  * surgical wound shows no sign of inflammation, or wound can be treated well in an outpatient setting
  * normal inflammatory markers (≤135 mg/l C-reactive protein (CRP), ≤9 10⁹/l white blood cell count)
Daily doses of analgetics | 30 days
  Amount, type, and time of application of analgetics will be obtained from medical and nursing records.
Postoperative pain | 7 days
  evaluated on the numeric rating scale (0 - 10, steps of 1)
Postoperative mobilization | 7 days
  Scoring:
  * 0: 24 h in bed
  * 1: Out of bed only to go to bathroom
  * 2: Out of bed on free will
Overall fluid intake | 7 days
  all fluids in ml per day
Blood pressure | 7 days
  3 times daily
Pulse | 7 days
  3 times daily (or more often if required)
Intensive care | 14 days
  number of days in intensive care unit
Well-being | 4 days
  well-being evaluating on day 2 and 4 after surgery using the Basle mental state scale as well as 5 additional items to evaluate the effects of caffeine. (Hobi 1985, Hobi 1989)
Sleep behaviour | 4 days
  Leeds Sleep Evaluation Questionnaire (LSEQ) on day 2 and 4 after surgery. (Parrott 1986)
Sleeping habits | 4 days
  Questionnaire evaluating duration and deepness of sleep.
Satisfaction with surgery | 4 days
  Questionnaire on day 4 about satisfaction of treatment
Consumption of sleep inducing drugs | 7 days
  amount and type of sleep inducing drugs

OTHER OUTCOMES:
preoperative caffeine consumption | before surgery
  Questionnaire evaluation the caffeine consumption of patients (type of beverages, amount etc)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Steffen, MD, Principal Investigator — Department of General, Visceral, Endocrine and Transplantation Surgery, Cantonal Hospital St. Gallen
Locations (2):
- Switzerland (2):
  - Department of General, Visceral, Endocrine and Transplantation Surgery, Cantonal Hospital St. Gallen, Rorschach
  - Department of General, Visceral, Endocrine and Transplantation Surgery, Cantonal Hospital St. Gallen, Sankt Gallen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muller SA, Rahbari NN, Schneider F, Warschkow R, Simon T, von Frankenberg M, Bork U, Weitz J, Schmied BM, Buchler MW. Randomized clinical trial on the effect of coffee on postoperative ileus following elective colectomy. Br J Surg. 2012 Nov;99(11):1530-8. doi: 10.1002/bjs.8885. Epub 2012 Sep 14. PMID 22987303
- [Background] Metcalf AM, Phillips SF, Zinsmeister AR, MacCarty RL, Beart RW, Wolff BG. Simplified assessment of segmental colonic transit. Gastroenterology. 1987 Jan;92(1):40-7. doi: 10.1016/0016-5085(87)90837-7. PMID 3023168
- [Background] Hobi V, Gerhard U, Gutzwiller F. [A report on experiences using Goldberg's GHQ (General Health Questionnaire)]. Schweiz Rundsch Med Prax. 1989 Feb 28;78(9):219-25. German. PMID 2928619
- [Background] Hobi V. Basler Befindlichkeits-Skala. Ein Self-Rating zur Verlaufsmessung der Befindlichkeit. Manual. 1 ed. Weinheim: Beltz Test GmbH, 1985.
- [Background] Parrott AC, Hindmarch I. The Leeds Sleep Evaluation Questionnaire in psychopharmacological investigations - a review. Psychopharmacology (Berl). 1980;71(2):173-9. doi: 10.1007/BF00434408. PMID 6777817
- [Derived] Abbassi F, Muller SA, Steffen T, Schmied BM, Warschkow R, Beutner U, Tarantino I. Caffeine for intestinal transit after laparoscopic colectomy: randomized clinical trial (CaCo trial). Br J Surg. 2022 Nov 22;109(12):1216-1223. doi: 10.1093/bjs/znac265. PMID 35909263
- [Derived] Kruse C, Muller SA, Warschkow R, Luthi C, Brunner W, Marti L, Sulz MC, Schmied BM, Tarantino I, Beutner U. Does caffeine reduce postoperative bowel paralysis after elective laparoscopic colectomy? (CaCo trial): study protocol for a randomized controlled trial. Trials. 2016 Apr 4;17:186. doi: 10.1186/s13063-016-1297-1. PMID 27044596
- See also: Web site of the Department of General, Visceral, Endocrine and Transplantation Surgery, Cantonal Hospital St. Gallen (German only) — http://www.chirurgie.kssg.ch/